CLINICAL TRIAL: NCT04375605
Title: RACE-trial: Neoadjuvant Radiochemotherapy Versus Chemotherapy for Patients With Locally Advanced, Potentially Resectable Adenocarcinoma of the Gastroesophageal Junction (GEJ) A Randomized Phase III Joint Study of the AIO, ARO and DGAV
Brief Title: Neoadjuvant RCT Versus CT for Patients With Locally Advanced, Potentially Resectable Adenocarcinoma of the GEJ
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other); Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Ralf Hofheinz, Prof. Dr. med., Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RACE; 2018-001728-20 (EudraCT Number); AIO-STO-0118 (Other: Arbeitsgemeinschaft Internistische Onkologie); 2024-516271-32-00 (EU CTIS Number)
Record Dates: First submitted 2020-04-21; First posted 2020-05-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (control arm) (Active Comparator): Patients randomized in control arm A will receive four cycles of neoadjuvant chemotherapy with FLOT every two weeks (5-FU 2600 mg/m² d1, folinc acid 200 mg/m² d1, oxaliplatin 85 mg/m² d1, docetaxel 50 mg/m² d1) followed by surgical resection 4-6 weeks after day 1 of the last cycle of neoadjuvant therapy. 6-12 weeks after surgery adjuvant chemotherapy starts with 4 cycles of FLOT (total treatment period 25-32 weeks).
  Interventions: Drug: 5-Fluorouracil; Drug: Calcium folinate; Drug: Oxaliplatin; Drug: Docetaxel
- Arm B (experimental arm) (Experimental): Patients randomized in experimental arm B will receive two cycles of neoadjuvant induction chemotherapy with FLOT (5-FU 2600 mg/m² d1, folinic acid 200 mg/m² d1, oxaliplatin 85 mg/m² d1, docetaxel 50 mg/m² d1) every two weeks (4 weeks of therapy) followed by radiochemo-therapy beginning at day 21 after day one of the last cycle of chemotherapy. Radiochemotherapy consists of oxaliplatin 45 mg/m² weekly (d1, 8, 15, 22, 29) and continuous infusional 5-FU 225 mg/m² plus concurrent radiotherapy given in 5/week fractions with 1.8 Gy to a dose of 45 Gy over 5 weeks. Resection is performed 4-6 weeks after last treatment with chemotherapy / radiation. Adjuvant treatment starts 6-12 weeks after surgery and consists of 4 cycles of FLOT (total treatment period of 26 - 33 weeks).
  Interventions: Drug: 5-Fluorouracil; Drug: Calcium folinate; Drug: Oxaliplatin; Drug: Docetaxel; Radiation: Radiation; Drug: Oxaliplatin during radiotherapy; Drug: 5-Fluorouracil during radiotherapy

INTERVENTIONS:
Drug: 5-Fluorouracil — Day 1 q2w: 2600 mg/m² IV over 24 hours
Drug: Calcium folinate — Day 1 q2w: 200 mg/m² IV over 2 hours
  Other Names: Folinic Acid
Drug: Oxaliplatin — Day 1 q2w: 85 mg/m² IV over 2 hours
Drug: Docetaxel — Day 1 q2w: 50 mg/m² IV over 2 hours
Radiation: Radiation — 25 fractions (5 each week over 5 weeks) each 1,8 Gy to a total of 45 Gy
  Arms: Arm B (experimental arm)
Drug: Oxaliplatin during radiotherapy — Day 1, 8, 15, 22, 29: 45 mg/m² IV over 2 hours
  Arms: Arm B (experimental arm)
Drug: 5-Fluorouracil during radiotherapy — day 1 - 33: 225 mg/m²/day IV continuously
  Arms: Arm B (experimental arm)

SUMMARY:
This is a multicenter, prospective, randomized, stratified, controlled, open-label study comparing neoadjuvant radiochemotherapy with FLOT versus FLOT chemotherapy alone für patients with locally advanced, potentially resectable adenocarcinoma of the gastroesophageal junction (GEJ)

DETAILED DESCRIPTION:
The RACE trial seeks to demonstrate superiority of preoperative FLOT induction chemotherapy followed by preoperative radiochemotherapy and postoperative FLOT chemotherapy over perioperative FLOT chemotherapy without radiotherapy in patients with adenocarcinoma of the gastroesophageal junction undergoing adequate oncological surgery.

Eligible patients will be randomly allocated to one of two treatment groups, i.e. preoperative chemotherapy (Arm A) or preoperative chemotherapy with subsequent preoperative radiochemotherapy (arm B), both followed by resection and postoperative completion of chemotherapy. Randomization will occur in a 1:1 ratio with stratification by primary tumor site (Siewert I vs. Siewert II/III).

Arm A:

Patients randomized to Arm A (control arm) will be treated with four preoperative cycles of FLOT. Cycles will be repeated every two weeks. The preoperative chemotherapy duration in Arm A is eight weeks. Surgical resection will follow 4-6 weeks after day 1 of the last cycle of neoadjuvant therapy. Postoperative chemotherapy will start 6-12 weeks after surgery and consists of another four cycles of FLOT every two weeks. The total treatment period is 25-32 weeks.

Arm B:

Patients randomized in Arm B (experimental arm) will be treated with two cycles of FLOT every two weeks. Radiochemotherapy will start three weeks after day 1 of the second cycle and consists of oxaliplatin and infusional 5-fluorouracil plus concurrent radiotherapy given to a dose of 45 Gy (25 daily fractions with 1.8 Gy) over five weeks. The preoperative treatment duration is 10 weeks. Surgical resection will follow 4-6 weeks after last treatment with chemotherapy / radiation. Postoperative chemotherapy will start 6-12 weeks after surgery and consists of four cycles of FLOT every two weeks. The total treatment period is 26-33 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven, locally advanced and potentially resectable adenocarcinoma of the gastroesophageal junction (GEJ) (Siewert I- III) that is: cT3-4, any N, M0 or cT2 N+, M0 according to AJCC 8th edition
2. Patients* must be candidates for potential curative resection as determined by the treating surgeon
3. ECOG performance status 0-1
4. Age 18 years or above
5. Adequate hematologic function with absolute neutrophil count (ANC) ≥ 1.5 x 10^9/l, platelets ≥ 100 x 10^9/l and hemoglobin ≥ 9.0 mg/dl
6. INR <1.5 and aPTT<1.5 x upper limit of normal (ULN) within 7 days prior to randomization
7. Adequate liver function as measured by serum transaminases (ASAT, ALAT) ≤ 2.5 x ULN and total bilirubin ≤ 1.5 x ULN
8. Adequate renal function with serum creatinine ≤ 1.5 x ULN
9. QTc interval (Bazett*) ≤ 440 ms
10. Written informed consent obtained before randomization
11. Negative pregnancy test for women of childbearing potential within 7 days of commencing study treatment. Males and females of reproductive potential must agree to practice highly effective*** contraceptive measures during the study and for 6 months after the end of study treatment. Male patients must also agree to refrain from father a child during treatment and up to 6 months afterwards and additionally to use a condom during treatment period. Their female partner of childbearing potential must also agree to use an adequate contraceptive measure.

    * *There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.
    * ** formula for QTc interval calculation (Bazett): QTc= ((QT) ̅" (ms)" )/√(RR (sec))= ((QT) ̅" (ms)" )/√(60/(Frequence (1/min)))
    * *** highly effective (i.e. failure rate of <1% per year when used consistently and correctly) methods: intravaginal and transdermal combined (estrogen and progestogen containing) hormonal contraception; injectable and implantable progestogen-only hormonal contraception; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence (complete abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments).

Exclusion Criteria:

1. Evidence of metastatic disease (exclusion of distant metastasis by CT of thorax and abdomen, bone scan or MRI [if osseous lesions are suspected due to clinical signs])
2. Past or current history (within the last 5 years prior to treatment start) of other malignancies. Patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible
3. Evidence of peripheral sensory neuropathy > grade 1 according to CTCAE version 4.03
4. Patients with other significant underlying medical conditions that may be aggravated by the study treatment or are not controlled
5. Pregnant or lactating females
6. Patients medically unfit for chemotherapy and radiotherapy
7. Patients receiving any immunotherapy, cytotoxic chemotherapy or radiotherapy other than defined by the protocol. The participation in another clinical trial with the use of investigational agents, chemotherapy or radiotherapy during the trial is not permitted
8. Known hypersensitivity against 5-FU, folinc acid, oxaliplatin or docetaxel
9. Other known contraindications against 5-FU, folinic acid, oxaliplatin, or docetaxel
10. Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, NYHA III-IV
11. Clinically significant valvular defect
12. Other severe internal disease or acute infection
13. Peripheral polyneuropathy > NCI Grade II according to CTCAE version 4.03
14. Chronic inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of PFS between arms | up to 5 years
  to compare PFS in patients with resectable GEJ adenocarcinoma receiving perioperative FLOT alone versus perioperative FLOT combined with neoadjuvant radiochemotherapy where PFS ist defined as the time from randomization to disease progression or disease recurrence after surgery or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  Overall survival (OS) where OS is defined as the time from randomization to death from any cause
R0 resection rate | after surgery, approx. 12 weeks after randomization
  R0 resection rate where R0 resection is defined as microscopically margin negative resection with no gross or microscopic tumor remains in the areas of the primary tumor and/or samples regianal lymph nodes based on evaluation by the local pathologist.
Number of harvested lymph nodes | after surgery, approx. 12 weeks after randomization
  Number of harvested lymph nodes during surgery
Site of tumor relapse | 5 years
  Site of tumor relapse if tumor recurrence/relapse occurs
Overall survival rate at 1, 3 and 5 years | 1 year, 3 years, 5 years
  Overall survival rate is defined as the proportion of patients known to be alive at 1, 3 or 5 years after randomization
Patient reported outcomes: quality of life according to questionnaire EORTC-QLQ-C30 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 68 months
  quality of life scores according to validated questionnaires EORTC-QLQ-C30
Patient reported outcomes: quality of life according to questionnaire EORTC module OG25 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 68 months
  quality of life scores according to validated questionnaire EORTC module OG25

CONTACTS AND LOCATIONS:
Overall Officials: Ralf-Dieter Hofheinz, Prof. Dr., Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Unversity Hospital Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenzen S, Biederstadt A, Ronellenfitsch U, Reissfelder C, Monig S, Wenz F, Pauligk C, Walker M, Al-Batran SE, Haller B, Hofheinz RD. RACE-trial: neoadjuvant radiochemotherapy versus chemotherapy for patients with locally advanced, potentially resectable adenocarcinoma of the gastroesophageal junction - a randomized phase III joint study of the AIO, ARO and DGAV. BMC Cancer. 2020 Sep 15;20(1):886. doi: 10.1186/s12885-020-07388-x. PMID 32933498